CLINICAL TRIAL: NCT05994443
Title: Fetal Brain Growth: Effects of Antenatal Corticosteroids on Fetal and Neonatal Brain Development - a Pilot Study
Brief Title: Fetal Brain Growth - Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: McGill University (Other); University of Arizona (Other)
Responsible Party: Principal Investigator, Jarred Garfinkle, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2023-8114
Record Dates: First submitted 2023-05-23; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Preterm Labor; Maternal Psychological Distress
Keywords: Antenatal corticosteroids; fetal brain growth
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women exposed to threatened preterm labor and exposed to antenatal corticosteroids: Pregnant women with threatened preterm labor (TPTL) who received antenatal corticosteroids (ACS) between 22 and 34 weeks and 6 days of gestation at our hospital.
- Non-exposed pregnant women: Pregnant women with normal pregnancies.

SUMMARY:
The goal of this observational prospective study is to explore the feasibility of measuring fetal and neonatal brain growth using 2D and 3D ultrasound in fetuses exposed to threatened preterm labor (TPTL) and antenatal corticosteroids (ACS) compared to non-exposed fetuses.

Patients with singleton pregnancies on our site with repeated ultrasound measurements every 4 weeks will be evaluated for fetal brain development. The exposed group is defined as patients with a dual exposure of TPTL and ACS. The non-exposed group will be composed of patients who did not have TPTL and ACS. Therefore, patients will have a maximum of 5 additional visits (4 that will occur prenatally and 1 postnatal visit).

DETAILED DESCRIPTION:
The investigators propose a monocentric prospective pilot cohort study of patients with singleton pregnancies admitted to the McGill University Health Centre (MUHC) - Royal Victoria Hospital (RVH) site with repeated ultrasound measurements every 4 weeks to evaluate fetal brain development. The exposed group is defined as patients with a dual exposure of TPTL and ACS. The non-exposed group will be composed of patients who did not have TPTL and ACS. Therefore, patients will have a maximum of 5 additional visits (4 that will occur prenatally and 1 postnatal visit). The investigators plan to recruit women over a period of 24 months and will need an additional period of 6 months to complete data extraction from delivery and perform all postnatal measures.

Primary Outcome: Our primary outcome will be the feasibility of a prospective observational study measuring fetal and neonatal brain growth using 2D and 3D ultrasound in fetuses exposed to TPTL and ACS to non-exposed fetuses. Feasibility will be defined on the following criteria: 1. Number of patients recruited per month; 2. Ability to recruit eligible patients and 3. Ability to successfully complete the 2D measures and 3D volumes for each ultrasound exam. Success will be defined by the following criteria: 1. At least two patients will be recruited per month; 2. At least 50% of all eligible patients exposed to TPTL and ACS will be recruited; 3. At least 50% of all 2D measures and 3D volumes could be obtained.

Secondary Outcomes: Our secondary outcomes will include 2D and 3D ultrasound measurements of fetal brain structures, more specifically: biparietal diameter, head circumference, corpus callosum length, corpus callosum-fastigium length, ventricular width, total fetal brain volume, frontal lobe volume, cerebellar volume, and thalamic volume (all measurements in cm). Neonatal brain structures will also be measured by 2D ultrasound, including corpus callosum length and corpus callosum-fastigium length (in cm).

Exposed patients will have a fetal ultrasound performed by a trained and qualified ultrasound technologist or a Maternal-Fetal Medicine specialist within 4 days of their admission to the hospital. Psychometric questionnaires will be filled on the same day. Ultrasounds will subsequently be performed at fixed gestational age: 24, 28, 32, and 36 weeks (+/- 4 days).

Non-exposed patients will have fetal ultrasound performed by a trained and qualified ultrasound technologist or a Maternal-Fetal Medicine specialist at 24, 28, 32, and 36 weeks (+/- 4 days). Psychometric questionnaires will be filled on each of those days.

ELIGIBILITY:
Inclusion Criteria:

Exposed group - TPL and ACS:

* 22-34 weeks and 6 days gestation at time of recruitment.
* Threatened preterm labor (TPTL)
* Administration of a partial or full course of ACS.
* Admission to the MUHC-RVH birthing center or the antenatal floor (D6S).
* Delivery planned at the MUHC-RVH or an institution around the Greater Montreal Area.

Non-exposed group:

* At or prior to 22 weeks gestation at time of recruitment.
* Delivery planned at the MUHC-RVH.

Exclusion Criteria:

* Major congenital anomalies, suspected fetal syndrome or genetic disease, or intra-uterine fetal growth restriction.
* Significant maternal disease which may cause preterm delivery or fetal growth restriction (e.g., severe infection, uncontrolled hypertension or diabetes).
* Patients who received more than one course of ACS prior to enrollment.
* Patients on any oral or other systemic corticosteroids, with the exception of inhaled corticosteroids.
* BMI over 35.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with singleton pregnancies on our site.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility - It is this a feasible project? | 2 years
  Our primary outcome will be the feasibility of a prospective observational study measuring fetal and neonatal brain growth using 2D and 3D ultrasound in fetuses exposed to TPTL and ACS to non-exposed fetuses. Feasibility will be defined on the following criteria: 1. Number of patients recruited per month; 2. Ability to recruit eligible patients and 3. Ability to successfully complete the 2D measures and 3D volumes (in cm) for each ultrasound exam. Success will be defined by the following criteria: 1. At least two patients will be recruited per month; 2. At least 50% of all eligible patients exposed to TPTL and ACS will be recruited; 3. At least 50% of all 2D measures and 3D volumes could be obtained (in cm).

SECONDARY OUTCOMES:
Prenatal ultrasound measurements | 2 years
  Our secondary outcomes will include 2D and 3D ultrasound measurements (in cm) of fetal brain structures, more specifically: biparietal diameter, head circumference, corpus callosum length, corpus callosum-fastigium length, ventricular width, total fetal brain volume, frontal lobe volume, cerebellar volume, and thalamic volume (all measurements in cm). Neonatal brain structures will also be measured by 2D ultrasound, including corpus callosum length and corpus callosum-fastigium length (in cm)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Maude Morency, MD, Principal Investigator — RI-MUHC
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be kept between collaborators.